CLINICAL TRIAL: NCT01628211
Title: Randomized Phase 2 Study Comparing Second Look Laparoscopy to Standard Follow up in Patients With no Radiologic Evidence of Disease at 6 Months After Complete Resection of Colorectal Mucinous Carcinoma
Brief Title: Second Look Laparoscopy in Colorectal Cancer
Acronym: HIPEC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC
Record Dates: First submitted 2012-06-20; First posted 2012-06-26 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
Keywords: hyperthermic chemotherapy; intraperitoneal chemotherapy; second-look laparoscopy; peritoneal carcinosis; mucinous colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Laparoscopy; Leucovorin; Fluorouracil; Oxaliplatin; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Second look laparoscopy (Experimental): Second look laparoscopy to evaluate for and treat peritoneal carcinosis
  Interventions: Procedure: Laparoscopy; Procedure: peritonectomy; Drug: Folinic Acid; Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: systemic chemotherapy
- standard follow up (No Intervention)

INTERVENTIONS:
Procedure: Laparoscopy — second look laparoscopy to evaluate for peritoneal carcinosis
  Arms: Second look laparoscopy
Procedure: peritonectomy — for patients with PCI < 20
  Arms: Second look laparoscopy
Drug: Folinic Acid — 20 mg/m2 IV given just before HIPEC for patients with PCI < 20
  Arms: Second look laparoscopy
Drug: 5-Fluorouracil — 400 mg/m2 IV given just before HIPEC in patients with PCI < 20
  Arms: Second look laparoscopy
Drug: Oxaliplatin — 460 mg/m2 intraperitoneal hyperthermic perfusion for patients with PCI < 20
  Arms: Second look laparoscopy
Drug: systemic chemotherapy — according to national Italian (AIOM) guidelines and may include biotherapies for patients with PCI > 20
  Arms: Second look laparoscopy

SUMMARY:
The purpose of this study is to evaluate whether a second-look laparoscopy, followed by peritonectomy, hyperthermic intraperitoneal chemotherapy (HIPEC) or systemic chemotherapy in case of peritoneal carcinosis, improves the overall survival of patients who have had radical resection of mucinous colorectal cancer.

DETAILED DESCRIPTION:
Patients will be entered into the study after radical resection of mucinous colorectal cancer, and reevaluated by CT scan after 6 months. Patients with no evidence of disease will be randomized to receive either standard follow up, or to have a second look laparoscopy to evaluate for peritoneal carcinosis. After laparoscopy, those patients who do not have peritoneal carcinosis will continue with standard follow up. Patients with peritoneal carcinosis diagnosed by laparoscopy will be treated according to their peritoneal carcinosis index (PCI). For patients with PCI > 20, systemic chemotherapy will be given according to Italian Association of Medical Oncology (AIOM) guidelines. Patients with PCI < 20 will undergo peritonectomy and then receive intravenous chemotherapy immediately followed by HIPEC.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis colorectal adenocarcinoma
* Mucinous histotype
* Stage I-III
* Radical (R0) surgical resection of primary tumor
* CT scan with contrast showing no evidence of disease recurrence 6 months after primary surgery
* Age ≥ 18 ≤ 65 years
* Performance Status ECOG ≤1
* Normal hepatic, renal and hematologic function
* Adjuvant chemotherapy permitted
* Signed informed consent

Exclusion Criteria:

* Residual disease after surgical resection of primary tumor
* Distant metastasis
* Active systemic infection
* Chronic cardiovascular illness that would contraindicate abdominal dilatation with pneumoperitoneum
* Concomitant or previous malignancy with 5 years of surgical resection of primary tumor (except for adequately treated non-melanoma skin cancer and in situ cervical cancer)
* Pregnancy or lactation
* Refusal or incapability of providing informed consent
* Impossibility of complying with study schedules and follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-04; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | two years

SECONDARY OUTCOMES:
number of patients with peritoneal carcinosis diagnosed at laparoscopy in the experimental arm | 6 months
changes in quality of life | 6 months
  quality of life is measured at baseline and 6 months after randomization
overall survival | five years
worst grade adverse event per patient | 7 months
  toxicity measured only in experimental arm, weekly from randomization to 30 days after experimental treatment
number of patients with radiologic evidence of disease after initial surgery | 6 months
list of therapies and clinical outcomes of patients who had radiologic evidence of disease within 6 months after initial surgery | two years
  description of therapies and outcomes for those patients who were not randomized due to presence of disease

CONTACTS AND LOCATIONS:
Overall Officials: C. Sassaroli, M.D., Principal Investigator — National Cancer Institute, Naples; A Cassata, M.D., Principal Investigator — University of Campania Luigi Vanvitelli; M.C. Piccirillo, M.D., Principal Investigator — NCI Naples
Locations (1):
- Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Entero-proctologico, Napoli, Italy